CLINICAL TRIAL: NCT03521089
Title: Cathodal Transcranial Direct Current Stimulation (tDCS) in Mild Cognitive Impairment (MCI): A Randomized, Double-Blind, Sham-Controlled Pilot Study
Brief Title: Cathodal tDCS in MCI: A Randomized, Double-Blind, Sham-Controlled Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yonas E Geda, MD, Professor of Neurology and Psychiatry, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-007478
Record Dates: First submitted 2018-03-29; First posted 2018-05-11 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment; Neurocognitive Dysfunction
Keywords: Mild Cognitive Impairment (MCI); Transcranial Direct Current Stimulation (tDCS)
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to active or sham transcranial direct current stimulation (tDCS) intervention
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tDCS (Active Comparator): Active tDCS uses the Soterix Medical 1x1 Low Intensity Transcranial Electrical Stimulator (tES) Model 2001. The active tDCS intervention include stimulation for 15 minutes at 1mA. The cathode electrode will be placed over the right dorsolateral prefrontal cortex with reference electrode (anode) over the left dorsolateral prefrontal cortex. Both electrodes are covered by saline-soaked sponges that are held against the scalp by a pair of large, adjustable head straps. Treatment sessions will last for 15 minutes. 5 consecutive treatment sessions will be completed within 1 week.
  Interventions: Device: Soterix Medical 1x1 Low Intensity Transcranial Electrical Stimulator (tES) Model 2001
- Sham tDCS (Sham Comparator): Sham tDCS uses the Soterix Medical 1x1 Low Intensity Transcranial Electrical Stimulator (tES) Model 2001. The sham tDCS intervention lasts for 15 minutes. The cathode electrode will be placed over the right dorsolateral prefrontal cortex with reference electrode (anode) over the left dorsolateral prefrontal cortex. Both electrodes are covered by saline-soaked sponges that are held against the scalp by a pair of large, adjustable head straps. Treatment sessions will last for 15 minutes. 5 consecutive treatment sessions will be completed within 1 week.
  Interventions: Device: Soterix Medical 1x1 Low Intensity Transcranial Electrical Stimulator (tES) Model 2001

INTERVENTIONS:
Device: Soterix Medical 1x1 Low Intensity Transcranial Electrical Stimulator (tES) Model 2001 — Transcranial direct current stimulation works by sending constant, low direct current through the electrodes. When these electrodes are placed in the region of interest, the current induces intracerebral current flow. This current flow then either increases or decreases the neuronal excitability in the specific area being stimulated based on which type of stimulation is being used. This change of neuronal excitability leads to alteration of brain function, which can be used in various therapies as well as to provide more information about the functioning of the human brain.
  Other Names: Soterix tDCS; Transcranial direct current stimulation; Non-invasive brain stimulation; Cathodal tDCS

SUMMARY:
This study evaluates the application of non-invasive brain stimulation in the treatment of Mild Cognitive Impairment (MCI) in adults aged 55-85. Half of the participants will receive transcranial direct current stimulation (tDCS), while the other half will receive sham (like placebo) stimulation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether giving transcranial direct current stimulation (tDCS) treatment using an investigational device called the Soterix tES Device (tDCS device) on the right side of the brain can improve performance on cognitive tests. Investigational means that the tDCS device is not approved by the U.S. Food and Drug Administration (FDA) for the use in this study.

tDCS is a non-invasive way to electrically stimulate the brain. The tDCS device is portable and runs on two 9-volt batteries. Electrodes from the tDCS device carry weak electrical current through the scalp and skull and into the brain. When the direction of the electric current flow is called cathodal, the brain under the site of stimulation reduces its activity.

When tasks are performed, certain parts of the brain are activated. Research studies have shown that younger adults and older adults activate similar parts of the brain when performing the same task (a memory task, for example). However, other researchers found older adults who scored worse on memory tasks, and those with Mild Cognitive Impairment, activated an additional part of the brain so both sides of the brain are activated. Researchers are not sure whether this additional activation is helpful or not. Investigators in this study believe that this extra activation may be contributing to worse performance on tasks.

It may be possible to use tDCS to reduce the brain activity on the extra activation (right) side in older adults, to resemble an activation pattern seen in younger adults (or higher scoring cohort). Using cathodal tDCS to reduce brain activity might help the brain in performing tasks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with confirmed MCI diagnosis
* Age 55-85
* Right handed (tested using the Edinburgh handedness inventory)
* Total PHQ-8 of ≤ 16 which signifies no severe depression
* All participants and/or caregivers must be able to provide informed consent

Exclusion Criteria:

* Neurodegenerative disease (e.g. Parkinson's, Huntington's, Multiple Sclerosis) other than MCI
* Previous brain lesion
* Intracranial abnormality such as prior stroke
* History of seizure disorder or epilepsy
* A "true" positive response, after patient clarification, to any question on the modified TMS/tDCS Adult Safety Screen questionnaire that would impact patient safety
* Any history of brain stimulation treatment (e.g., electroconvulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), vagal nerve therapy (VNS), deep brain stimulation (DBS))
* Use of any investigational drug within 4 weeks
* Cardiac pacemakers, implanted medication pumps, intracardiac lines; acute or unstable cardiac disease; intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head (exception: mouth/dental work) that cannot be safely removed
* Known or suspected pregnancy (extremely unlikely as the age range for this study is 55-85 years)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yonas E Geda, MD, MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (5.7) | 70.0 (9.5) | 70.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Flanker Inhibitory Control and Attention Test Scores
Description: Post-intervention score comparison between the intervention and control group measured by the NIH Toolbox Cognition Battery Test. The NIH Toolbox Cognition Battery Test is a comprehensive set of neuro behavioral measurements used to assess cognitive, sensory and motor functions where a higher composite score equals better cognitive performance. The NIH Toolbox Cognitive Scores used the Fully Adjusted Scale score (also referred to as the fully corrected T-score) with a mean of 50 and standard deviation of 10.
Time Frame: Baseline, 1-month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 35.1 (1.3) | 41.5 (1.3)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.0039, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.0156, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Picture Vocabulary Test Scores
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 52.0 (1.2) | 52.0 (1.2)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.9674, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.0938, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.2500, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in List Sorting Working Memory Test Scores
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 60.5 (1.9) | 51.8 (1.9)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.0067, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.0313, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.7500, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Dimensional Change Card Sort Test
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 43.7 (2.8) | 48.0 (2.8)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.3069, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.1875, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.7188, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change in Pattern Comparison Processing Speed Test Scores
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 46.6 (3.0) | 51.6 (3.0)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.2609, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.0313, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.0156, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change in Picture Sequence Memory Test v2.1 Score
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 45.2 (3.8) | 42.8 (3.8)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.6951, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.0938, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 0.0938, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Change in Oral Reading Recognition Test Score
Description: as for outcome 1
Time Frame: Baseline, 1 month post intervention
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 8 | 8
score on a scale | 58.5 (1.7) | 56.1 (1.7)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; Test type: Superiority; p = 0.3592, ANCOVA
Statistical Analysis 2: Comparison: Active tDCS; Test type: Superiority; p = 0.0625, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Sham tDCS; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: A symptom-based questionnaire was used to measure adverse events and was administered at each intervention visit for the 5 consecutive days over a total study duration of 12 months.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03521089/Prot_SAP_000.pdf